CLINICAL TRIAL: NCT05057221
Title: A Pilot Study to Assess the Safety, Tolerability and Efficacy of Selectin Inhibitor Uproleselan (GMI-1271) in Patients With COVID-19 Pneumonia
Brief Title: Safety, Tolerability and Efficacy of Uproleselan (GMI-1271) in Patients With COVID-19 Pneumonia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No more eligible patients were available.
Sponsor: Lena Napolitano, MD (Other)
Collaborators: GlycoMimetics Incorporated (Industry)
Responsible Party: Sponsor-Investigator, Lena Napolitano, MD, Medical Director and Professor of Surgery, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00195034
Record Dates: First submitted 2021-09-23; First posted 2021-09-27 (Actual); Results first posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: COVID-19 Pneumonia
Keywords: Uproleselan; Selectin Inhibitor
MeSH Terms: interventions — uproleselan

STUDY DESIGN:
Intervention Model Description: This is a prospective, interventional, single-arm, open label trial, with 1:1 matched de-identified retrospective control cohort.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Uproleselan (Experimental): Uproleselan injection is a sterile solution for IV administration, supplied in single-dose vials at a concentration of 50 mg/mL.
  Interventions: Drug: Uproleselan

INTERVENTIONS:
Drug: Uproleselan — Uproleselan 20 mg/kg BID up to maximum dose of 2500 mg, infused IV over 20 minutes on days 1-7 or until hospital discharge. It should be administered intravenously (IV) into a peripheral line, a central catheter, or a peripherally inserted central line catheter (PICC). Infusion should take place at a steady rate over a period of 20 minutes ±2 minutes using a syringe pump or IV pump.

SUMMARY:
The purpose of this study is to find out whether the drug uproleselan can help patients with severe COVID-19 pneumonia. Investigators will study both the side effects of the drug and assess if the drug will help patients recover more quickly and slow down the progression of acute respiratory failure.

DETAILED DESCRIPTION:
Soluble E-selectin is a significant biomarker for adult respiratory distress syndrome (ARDS). Soluble E-selectin also has pro-inflammatory properties further releasing cytokines and promoting its synthesis and the continued influx of neutrophils. Small molecule glycomimetic antagonists of E-selectin (rivipansel and uproleselan) are 500- to 1000-fold more potent inhibitors of E-selectin and have shown activity and no measurable toxicity in human clinical trials for other indications. Treatment with these E-selectin inhibitors reduced the levels of soluble E-selectin in the bloodstream which occurs during recovery of ARDS. Thus, antagonists of E-selectin which include glycomimetic antagonists and more specifically, rivipansel (GMI-1070) and uproleselan (GMI-1271), may be used to treat COVID-19 patients with respiratory symptoms that may lead to ARDS

Primary Objective:

Safety of uproleselan in patients with severe COVID-19 pneumonia.

Secondary Objectives:

To evaluate if treatment with uproleselan administered intravenously in addition to the best available therapy according to institutional guidelines is able to reduce the progression of acute respiratory failure, in patients with severe COVID-19 pneumonia.

* To evaluate proportion of patients alive and free of respiratory failure through Day 28
* To evaluate overall survival and all-cause mortality at day 15 and 28.
* To evaluate changes in the COVID ordinal outcomes scale.
* To assess adverse events to evaluate the safety of uproleselan.
* To assess ventilator-free days, ICU-free days, oxygen, vasopressor free days.
* To evaluate changes in D-dimer.

Exploratory Objectives:

* To examine the correlation of plasma soluble E-selectin concentrations with clinical outcomes.
* To examine the correlations of other biomarkers of interest with clinical outcome.

Previous versions of this record mistakenly suggested the trial would assess the number of participants who experienced a Grade 3-5 hemorrhagic event. The outcome title has been corrected to state the number of participants with a Grade 3-4 hemorrhagic event were assessed, as the scale used does not go to Grade 5.

ELIGIBILITY:
Inclusion Criteria:

* Documented COVID-19 pneumonia: defined as upper respiratory tract specimen (nasopharyngeal swab (NPS) or viral throat swab) positive for COVID-19 and/or imaging at computed tomography scan suggestive of COVID-19 pneumonia.
* Confirmed coronavirus (SARS-CoV-2) (positive real-time reverse transcription polymerase chain reaction test (RT-PCR) for SARS-CoV-2 within 72 hours) enrolled ≤ 48 hours of need for supplemental oxygen.
* Currently hospitalized requiring supplemental oxygen.
* Have severe COVID-19 according to the World Health Organization (WHO) Interim Guidance with confirmation by real-time RT-PCR assay. The enrollment criteria with one of the following: respiratory distress, respiratory rate (RR) ≥30 beats/min; oxygen saturation level less than 93% in resting state; or partial pressure of oxygen (PaO2)/oxygen concentration (FiO2) ≤ 300 mmHg.
* Willing and able to participate in all required evaluations and procedures.

Exclusion Criteria:

* In the opinion of at least two investigators, unlikely to survive for >48 hours from screening.
* Severe chronic respiratory disease (e.g. Chronic obstructive pulmonary disease or other) requiring supplemental oxygen and/or having required mechanical ventilation pre-COVID-19 infection.
* Concurrent enrollment in a COVID related interventional drug trial. Use of remdesivir, steroids, and convalescent plasma are permitted along with other standard of care therapies for COVID.37
* Currently on invasive mechanical ventilation.
* Hypotension defined as systolic blood pressure < 90 mmHg on two sequential readings at least 4 hours apart.
* Total Bilirubin ≤ 3 x upper limit of normal (ULN), Creatinine Clearance ≥ 30 mL/min/1.73m2.
* Pregnant or breastfeeding.
* Known diagnosis of an acute thrombosis on admission.
* Concurrent dual antithrombotic therapy (aspirin or P2Y12 inhibitor plus anticoagulation to treat deep venous thrombosis or pulmonary embolism (single antiplatelet or anticoagulant agent at prophylactic dose is permitted).
* Concomitant use of thrombolytic therapy.
* Concomitant therapeutic systemic anticoagulant therapy (e.g. heparin, warfarin, direct thrombin inhibitors and direct factor Xa inhibitors). As per NIH Guidelines: Hospitalized adults with COVID-19 should receive Venous thromboembolism (VTE) prophylaxis per the standard of care for other hospitalized adults (AIII). Anticoagulant or antiplatelet therapy should not be used to prevent arterial thrombosis outside of the usual standard of care for patients without COVID-19 (AIII); https://www.covid19treatmentguidelines.nih.gov/therapeutic-management/
* History of recent major bleeding, defined in accordance with the criteria of the International Society on Thrombosis and Hemostasis (ISTH).
* History of bleeding disorder thought to impose excessive bleeding risk as per investigator discretion
* Hemodynamic instability, defined as inability to maintain mean arterial pressure.
* Hypersensitivity to the active substance or to any of the excipients of uproleselan.
* Any physical examination findings and/or history of any illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk to the patient by their participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lena Napolitano, MD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Uproleselan
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Adults with confirmed severe COVID-19 pneumonia (WHO definition) requiring supplemental oxygen
Arm/Group | Uproleselan
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6
Body Mass Index (BMI [Mean (Standard Deviation); unit: Kg/m^2] | 37.21 (10.36)
E-selectin Plasma Concentrations [Mean (Standard Deviation); unit: nanograms divided by milliliters] | 15.83 (6.479)

OUTCOME MEASURES:

1. Primary Outcome: Safety of Uproleselan - as Measured by Serious Adverse Events
Description: Descriptive statistics will be calculated for quantitative safety data
Time Frame: Up to 28 days
Measure: Number; unit: Serious Adverse Events
Arm/Group | Uproleselan
Number analyzed (Participants) | 6
Serious Adverse Events | 0

2. Primary Outcome: Safety of Uproleselan- as Measured by Frequency of Serious Adverse Events
Description: Frequency counts will be compiled for classification of qualitative safety data.
Time Frame: Up to 28 days
Measure: Number; unit: daily events
Arm/Group | Uproleselan
Number analyzed (Participants) | 6
daily events | 0

3. Secondary Outcome: Change in the Progression to Acute Respiratory Failure for Patients With a Baseline PaO2/FiO2 >= 200
Description: Patients with a baseline PaO2/FiO2 >= 200: progression of respiratory failure is defined by:
  1. severe gas transfer deficit (PaO2/FiO2 < 200);
  2. persistent respiratory distress while receiving oxygen (persistent marked dyspnea, use of accessory respiratory muscles, paradoxical respiratory movements); The rate will be calculated as the proportion of patients who experienced at least one of the events above by day+15 from treatment start.
Time Frame: Enrollment, 15 days
Measure: Count of Participants; unit: Participants
Arm/Group | Uproleselan
Number analyzed (Participants) | 6
Participants | 0

4. Secondary Outcome: Number of Patients Alive Who Are Free of Respiratory Failure
Description: Number of patients alive and free of acute respiratory failure which required initiation of mechanical ventilation
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Uproleselan
Number analyzed (Participants) | 6
Participants | 6

5. Secondary Outcome: All-cause Mortality
Description: All-cause hospital mortality
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Uproleselan
Number analyzed (Participants) | 6
Participants | 0

6. Secondary Outcome: Time to Change Oxygenation
Description: Number of days it took to reduce their oxygen requirements
Time Frame: during hospitalization; hospital stay ranged from 2 to 10 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Uproleselan
Number analyzed (Participants) | 6
Days | 2 (1)

7. Secondary Outcome: Number of Patients Requiring Mechanical Ventilation
Description: Number of patients requiring mechanical ventilation
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Uproleselan
Number analyzed (Participants) | 6
Participants | 0

8. Secondary Outcome: Change in the World Health Organization (WHO) COVID-19, "8-point Ordinal Scale" as Shown by Presenting Selected Time Points Through Day 28
Description: WHO COVID-19, "8-point ordinal scale" has a range of 1-8 with higher numbers indicating a more severe disease.
Time Frame: Enrollment, day 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Uproleselan
Number analyzed (Participants) | 6
score on a scale
  Day 1 | 4.67 (0.42)
  Day 3 | 2.8 (0.74)
  Day 15 | 1.17 (0.16)
  Day 28 | 1.20 (0.2)

9. Secondary Outcome: Actual Duration of Hospitalization
Description: Duration of hospitalization - number of inpatient hospital days. Participants were planned to be followed for up to 28 days, although the longest actual hospital stay for a participant was 10 days.
Time Frame: Up to 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Uproleselan
Number analyzed (Participants) | 6
days | 4.67 (2.56)

10. Secondary Outcome: Actual Duration of ICU Care
Description: Duration of ICU stay - number of ICU days. Participants were planned to be followed for up to 28 days, although the longest actual hospital stay for a participant was 10 days.
Time Frame: Up to 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Uproleselan
Number analyzed (Participants) | 6
days | 1.33 (1.89)

11. Secondary Outcome: Participants Who Experienced Grade 3-4 Hemorrhagic Events
Description: Number of participants who experienced a Grade 3 or Grade 4 hemorrhagic event based on the World Health Organization's (WHO) Bleeding Scale. On the scale, a Grade 3 event means gross blood loss, and a Grade 4 event means debilitating blood loss.
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Uproleselan
Number analyzed (Participants) | 6
Participants | 0

12. Secondary Outcome: Change in E-selectin Plasma Concentrations, as Shown by Values for Each of Those Days
Description: Changes in E-selectin plasma concentrations measured each day for 6 days.
Time Frame: 6 Days
Measure: Mean (Standard Deviation); unit: Nanograms divided by milliliter
Arm/Group | Uproleselan
Number analyzed (Participants) | 6
Nanograms divided by milliliter
  Day 1 | 19.19 (9.783)
  Day 2 | 15.15 (6.524)
  Day 3 | 18.15 (9.660)
  Day 4 | 18.09 (7.239)
  Day 5 | 27.04 (0.000)
  Day 6 | 26.85 (0.000)

13. Secondary Outcome: Participants Who Experienced Venous Thromboembolism (Deep Venous Thrombosis or Pulmonary Embolism)
Description: Venous thromboembolism - DVT or PE
Time Frame: Enrollment, up to day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Uproleselan
Number analyzed (Participants) | 6
Participants | 0

14. Secondary Outcome: Number of Mechanical Ventilation and Vasopressor Days
Description: Days of mechanical ventilation and days of vasopressors
Time Frame: Up to Day 28
Measure: Number; unit: days
Arm/Group | Uproleselan
Number analyzed (Participants) | 6
days
  Days of mechanical ventilation | 0
  vasopressor days | 0

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Uproleselan
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Uproleselan (N=6)
bilateral leg edema (Blood and lymphatic system disorders) | 1
dizziness (Ear and labyrinth disorders) | 1
mild diarrhea and indigestion (Gastrointestinal disorders) | 1
bruising from clinical blood draws (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT05057221/Prot_SAP_000.pdf